CLINICAL TRIAL: NCT04376931
Title: A Prospective Dose Finding Study of Iscador Infusion: Phase Ib Study With Prolonged Observation (ISINFULA)
Brief Title: A Prospective Dose Finding Study of Iscador Infusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISINFULA 37-04
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Advanced Cancer
Keywords: advanced malignant disease; mistletoe; Iscador

STUDY DESIGN:
Intervention Model Description: Prospective, dose-escalating mono-center open label dose-finding study without control group (3+3 design), including a follow-up on-treatment observation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iscador®P as intravenous infusion (Experimental): Investigational therapy will be administered in six Dose Groups (DG):
  10 mg, 20 mg, 40 mg, 90 mg, 140 mg and 200 mg Iscador®P. The initial dose group of the study is set to 40 mg Iscador®P. The two lower dose groups (20 or 10 mg) will only be used in case of intolerance at 40 mg Iscador®P. Once per week patients receive intravenous infusions of Iscador®P dissolved in 250 ml of sodium chloride solution (0.9 %). After the 4-week period of the MTD estimation phase each subject will immediately be included into a follow up observation in which he/she receives the last well tolerated dosage they had or the next lower dosage than the currently investigated DG in the running phase Ib study depending on the current estimate of the MTD at that time.
  Interventions: Drug: Intravenous Solution

INTERVENTIONS:
Drug: Intravenous Solution — Iscador®P: fermented aqueous extract of mistletoe grown on pine tree (Viscum album L. subspecies austriacum (Wiesb.) Vollmann), licensed for subcutaneous (SC) application in Switzerland, Germany, Austria, Sweden, and South Korea in dosages up to 20 mg.
  Other Names: ISINFULA

SUMMARY:
Prospective, dose-escalating mono-center open label dose-finding study without control group (3+3 design), including a follow-up on-treatment observation. In this study will be recruited 15 patients with a histologically or cytologically confirmed diagnosis of an advanced malignant disease during a therapy-free interval.Investigational drug:Iscador®P: fermented aqueous extract of mistletoe grown on pine tree (Viscum album L. subspecies austriacum (Wiesb.) Vollmann), licensed for subcutaneous (SC) application in Switzerland, Germany, Austria, Sweden, and South Korea in dosages up to 20 mg.

The initial dose group of the study is set to 40 mg Iscador®P.

DETAILED DESCRIPTION:
This is a prospective open label dose finding study (phase I) of Iscador®P in patients with histological or cytological confirmed diagnosis of an advanced malignant disease during a therapy-free interval. Primary objective : To determine the maximum tolerated dose (MTD) of Iscador®P as intravenous infusion in the aforementioned patient population, based on the incidence of dose-limiting toxicities (DLTs). Secondary objective :To investigate safety and tolerability of long-term intravenous infusion of Iscador®P based on incidence and severity of adverse drug reactions.

All patients are receiving best supportive care and may receive, if necessary, specified concomitant therapies, which should not interfere with the safety parameters chosen for this study.

Investigational therapy will be administered in six Dose Groups (DG): 10 mg, 20 mg, 40 mg, 90 mg, 140 mg and 200 mg Iscador®P. The initial dose group of the study is set to 40 mg Iscador®P.

The two lower dose groups (20 or 10 mg) will only be used in case of intolerance at 40 mg Iscador®P. Once per week patients receive intravenous infusions of Iscador®P dissolved in 250 ml of sodium chloride solution (0.9 %). After the 4-week period of the MTD estimation phase each subject will immediately be included into a follow up observation in which he/she receives the last well tolerated dosage they had or the next lower dosage than the currently investigated DG in the running phase Ib study depending on the current estimate of the MTD at that time.

Study entry of individual patients will be set apart by one week. Dosages of subsequent dose groups depend on the incidence of DLTs in former groups.

For safety reasons the values of endotoxin content in Iscador®P, measured by the limulus test, are considered as the real content of endotoxins although the mistletoe lectins are cross reacting in this test. This leads to a maximum dose of 200 mg representing the upper limit of this dose finding study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily given written informed consent.
* ≥18 years of age.
* Metastatic or locally advanced solid tumor, histologically or cytologically confirmed, no standard therapy available or standard therapy has failed.
* Adequate organ function
* Life expectancy ≥ 3 months, ECOG ≤ 2.
* No ongoing or preceding therapy with mistletoe products.
* Women of childbearing potential: negative serum pregnancy test at screening, use of two adequate barrier methods
* Compliance with protocol, legal competence.

Exclusion Criteria:

* - Systemic cytotoxic chemotherapy, biological therapy, radiation therapy, OR major surgery prior trial treatment.
* Persisting toxicity of NCI-CTCAE Grade >1 related to prior therapy (Sensory neuropathy of Grade ≤2 is acceptable).
* Expected to require any other form of systemic or localized antineoplastic therapy while on trial
* Systemic corticosteroid therapy received ≤ 3 days prior to trial treatment or other forms of systemic immunosuppressive medication (except corticosteroids against immune-related AEs and /or premedication for IV contrast allergies/reactions; corticosteroid replacement therapy)
* Tumor and/or metastases of the CNS and/or carcinomatous meningitis
* Active infection requiring intravenous systemic therapy, HIV, severe allergic illness (including asthma), active tuberculosis, inflammatory diseases with body temperature > 38° C.
* Known hypersensitivity to mistletoe products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Subjects will be in this study for up to 58 weeks ( 4 weeks of treatment and follow-up for a maximum of 52 weeks if subjects are deemed to have continuous clinical benefit from the Iscador®P infusions.
  Maximum tolerated dose (MTD) of Iscador®P infusions, i.e. the dose eliciting dose-limiting toxicities (DLTs) in a maximum of 1 out of 6 patients treated at that dose.treated at that dose.

SECONDARY OUTCOMES:
Quality of Life as Assessed Using Functional Assessment of Cancer Therapy - General (FACIT-G) | Baseline and prior to each infusion in phase I and monthly in the follow-up period.4 weeks and follow up period for a maximum of 52 weeks
  The FACIT-F evaluates quality of life using 5 categories: physical well-being (PWB), social/family well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and fatigue (FS). Participants answer each item on a 5-point scale from 0 to 4. The total score is the sum of individual responses across all 5 categories and may range from 0 to 160. The FACIT-General (FACIT-G; range 0 to 108) is the sum of scores for PWB, SWB, EWB, and FWB; the FACIT-Fatigue (FACIT-F) trial outcome index (TOI; range 0 to 108) is the sum of scores for PWB, FWB, and FS; and the FACIT-F fatigue (range 0 to 52) is the sum of scores for the FS only. For derivations of the FACIT-F reported here, higher scores indicate better quality of life. The mean score at each timepoint was determined by averaging scores among all participants.
Incidence of adverse drug reactions (ADRs). | Subjects will be in this study for up to 58 weeks ( 4 weeks of treatment and follow-up for a maximum of 52 weeks if subjects are deemed to have continuous clinical benefit from the Iscador®P infusions.
  frequency of ADRs to intravenous mistletoe treatment will be measured during the study.
Tumor response | 4 weeks and follow up period for a maximum of 52 weeks
  Evaluation of tumor response will be according to the RECIST criteria V1.1
Progression-free survival | 4 weeks and follow up period for a maximum of 52 weeks
  Time to disease progression will be defined as the time from first infusion of Iscador®P to the date of documentation of disease progression.
Overall survival | 4 weeks and follow up period for a maximum of 52 weeks
  Overall survival will be measured from the date of first infusion of Iscador®P until the date of the last follow-up or death.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Bar Sela, Prof, Principal Investigator — Haemek MC
Locations (1):
- Haemek MC, Afula, North, Israel

IPD SHARING:
Plan to Share IPD: No